CLINICAL TRIAL: NCT05230264
Title: Examination of Sex-specific Differences in the Stress Response to Abdominal Aortic Aneurysm Repair - A Prospective Cohort Study
Brief Title: Sex-specific Differences in the Stress Response to Abdominal Aortic Aneurysm Repair
Acronym: SSStressAAA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21SM7254
Record Dates: First submitted 2022-01-18; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Abdominal Aortic Aneurysm; Stress; Surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men: Elective AAA Repair
  Interventions: Other: Elective AAA Repair
- Women: Elective AAA Repair
  Interventions: Other: Elective AAA Repair

INTERVENTIONS:
Other: Elective AAA Repair — Elective AAA Repair - Observation of Stress Response

SUMMARY:
It is recognised that women are at greater risk of death, complications and longer hospital stay following intact abdominal aortic aneurysm (AAA) repair, and the reason for this is not yet established. This disparity in outcomes for women compared to men is also recognised in other forms of cardiovascular surgery, which raises the question of whether women and men are reacting differently to the stress of operative repair.

This study aims to examine whether there are differences baseline stress markers and in the stress response to AAA repair between men and women. It will also examine whether markers of stress are associated with poor clinical outcomes and slower recovery (indicated by longer hospital stay).

The study will take the form of an observational cohort study. It will not alter any of the treatment that men and women receive, but will monitor their stress levels using physiological markers (through ECG (electrocardiogram) monitoring using a non-invasive holter, biochemical markers using blood samples (which will be taken at the same time as routine testing, so as not to require further invasive procedures), and psychological testing, using short forms that the patient will be able to fill out independently at different stages of their recovery. Clinical data will be used to look for relevant factors (clinical history or medications) which may alter the stress markers we are observing, and to compare outcomes with markers of stress.

Patients will be asked for their consent to share their data with the research team in order to participate in the study. It will be made clear that there will be no change in their clinical or operative management if they participate in the study and they will be able to withdraw consent for further participation at any time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women undergoing primary elective intact AAA repair, open or endovascular (EVAR) at participating centres.
* Capacity to consent.

Exclusion Criteria:

* Participants undergoing a secondary or emergency aortic procedure, or procedure for alternative aortic pathology.
* Relevant confounding pathology such as hypothalamic-pituitary axis pathology (e.g. Addison's disease).
* Lack of capacity to consent.
* Participants with pacemaker dependency, or a significant arrhythmia, will be excluded from analysis of heart rate variability, but will be included in the study for analysis of psychological and biochemical markers of stress.
* Participants on steroid treatment will also be excluded from analysis of biochemical markers but may be included for analysis of physiological markers and/or heart rate variability.
* Participants must be over the age of 50 (In order to facilitate capture of degenerative aortic aneurysmal pathology rather than an alternative aortic pathology e.g. traumatic, connective tissue disorder).

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women undergoing primary elective intact AAA repair, open or endovascular (EVAR) at participating centres.
  Consecutive recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical measures of stress: level of serum cortisol & dehydroepiandrosterone (DHEA) | Samples taken on the morning of operation (baseline), at anaesthetic induction, at the end of the procedure, 6 hours post-procedure and early morning samples during the remaining inpatient stay.
  Sex-specific differences in baseline and timing/magnitude of response to operative stress.

SECONDARY OUTCOMES:
Physiological parameters: assessment of beat-to-beat heart rate variability metrics. | Baseline recording compared to post-operative recording of patient recovery during inpatient stay.
  Sex-specific differences in baseline and timing/magnitude of response to operative stress.
Psychological measures of stress: measured by State Trait Anxiety Inventory-Y and self assessment (Likert Scale). | Pre-operative assessment compared to post-operative assessment at specified intervals during operative recovery - 2, 14, 30 and 90 days post-operation.
  Sex-specific differences in the baseline and timing/magnitude of response to operative stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided